CLINICAL TRIAL: NCT00511251
Title: Analysis of Induced Sputum and Lung Biopsies by SEM: a Tool to Identify Source of Exposure of Workers to Hazardous Dust
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TASMC-07-LF-07226-CTIL
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2007-08-03 (Estimated); Status verified 2007-08

CONDITIONS: Occupational Exposed Population
Keywords: IS-SEM

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim : to validate the qualitative analysis by Scanning Electron Microscope (SEM) of lung samples first in induced sputum in correlation to disease second by comparing hazardous particles in induced sputum to the analysis in lung tissue and finally by assessing if the particles present in transplanted patients correlated with occupational history.

DETAILED DESCRIPTION:
Abstract

Background: On the last few years there is a rise in the public awareness of the danger potential that lies in the exposure to hazardous dust in different professions. The examination of induced sputum has been used from the early eighties to research and diagnose inflammatory lung diseases. We assess here patients with lung disease and occupational history, in order to undergo work up to assess hazardous dust exposure.

Aim : to validate the qualitative analysis by Scanning Electron Microscope (SEM) of lung samples first in induced sputum in correlation to disease second by comparing hazardous particles in induced sputum to the analysis in lung tissue and finally by assessing if the particles present in transplanted patients correlated with occupational history.

Methods: 40 patients referred with occupational history were included. For 24 of them SEM analysis was done in induced sputum (IS) together with questionnaires and in 11 among them the SEM analysis was done both from lung tissue (TS) and IS. In addition 11 lung biopsies from patients with occupational history were scanned by SEM and compared to 10 biopsies from patients with no occupational history.

ELIGIBILITY:
Inclusion Criteria:

* Occupational exposed workers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-01; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fireman Elizabeth, PhD, Principal Investigator — TASMC